CLINICAL TRIAL: NCT05137678
Title: The Safety and Effectiveness of Glibenclamide in the Treatment of Aneurysm Subarachnoid Hemorrhage（aSAH）: a Randomized Controlled Clinical Study
Brief Title: Evaluate the Use of Glibenclamide on Acute aSAH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Guangzhi Shi, chief physician, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: glibenclamide study group2
Record Dates: First submitted 2021-10-19; First posted 2021-11-30 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid hemorrhage; Brain aneurysms; Glibenclamide
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm | interventions — Glyburide

STUDY DESIGN:
Intervention Model Description: Patients in the case group were treated with glibenclamide within 10 hours after onset, orally or through nasogastric tube, 1.25 mg each time, once every 8 hours, for 7 consecutive days. The control group was blank control.
Masking Description: Open label, result blind method
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Glibenclamide was given orally or through nasogastric tube, 1.25 mg every 8 hours for 7 days
  Interventions: Drug: glibenclamide
- Control group (No Intervention): No glibenclamide treatment

INTERVENTIONS:
Drug: glibenclamide — Glibenclamide was given orally or by nasal feeding
  Other Names: Glebenzene
  Arms: Experimental group

SUMMARY:
A randomized, open-labeled, blank-controlled and prospective trial meant to evaluate the use of glibenclamide on acute aneurysmatic subarachnoid hemorrhage. Patients will allocated randomly in two groups, one for 3.75 mg daily intake of glibenclamide for 7 days and another as a blank contrast. General clinical data and late cognitive status will be accessed in both groups.

DETAILED DESCRIPTION:
The study is a open-labeled, blank-controlled, prospective and randomized clinical trial, conducted at Tiantan Hospital and Tongren Hospital, affiliated with the Capital Medical University. Patients will be recruited from intensive care units. Appropriate ethics and regulatory approvals will be sought for all subjects, according to the International Conference on Harmonization guidelines for good clinical practice (ICH GCP). Investigators will obtain informed written consent from all patients or their legal representative. Recruitment will take place between 2021 and 2022.

Patients will be randomly assigned (1:1) to receive either glibenclamide 3.75mg or blank contrast. A computer-generated randomization code will be used to randomize patients. Patients will start treatment as soon as possible within 48 h of the stroke, with a daily dose till the 7 days after the recruitment. Trial medication consisted of one and a half pieces of tablet a day, given orally or via a nasogastric tube. Aneurysm treatment, either by microsurgery or embolization, will be performed as soon as possible, according with the standard of care for the recruiting center. Nimodipine 60mg, every six hours, will be started on admission and continued till two weeks later, in all patients as standard of care.

Patient's demographics, medical history and relevant investigation results will be collected. The severity of the hemorrhage will be clinically assessed by World Federation of Neurosurgical Societies grading scale and radiologically using the modified Fischer scale. At 90 days of follow up patients will be interviewed with modified Rankin scale (mRS) questionnaire (a scale that measures degree of incapacity/ dependence and mortality after neurological events) by a physician with no knowledge of treatment allocation. The main hypothesis is that, once compared with standard of care, glibenclamide 3.75mg will provide better clinical outcome and additionally will decrease mortality and improve quality of life and cognitive performance after 90 days.

Sample size: Previous studies have shown that the NSE mean for the third day after subarachnoid hemorrhage is 21 ng/ml, the standard deviation is about 3 ng/ml, and the third day NSE in patients with a good prognosis group is about 19 ng/ml, and the standard deviation is about 3 ng/ml; according to the two-sided test, significance of 5%, two groups of equal number of people, 90% of the degree of certainty, the calculation of the sample size of 98 cases, assuming 10% of the loss of visits, the total sample size is expected to be 110 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Subarachnoid hemorrhage was diagnosed by digital subtraction angiography, computed tomographic angiogram or magnetic resonance angiography;
2. Within 48 hours;
3. Age > 18 years old;
4. The expected length of stay is more than 7 days;
5. Sign informed consent.

Exclusion Criteria:

1. There was a history of taking sulfonylureas within 30 days before brain injury;
2. Combined with neurological or mental diseases, including stroke, epilepsy and dementia;
3. Hunt & Hess grade V patients;
4. Severe brain injury (central hernia or hook hernia within 48 hours after admission or after resuscitation) that cannot be solved at present;
5. History of alcohol or illicit drug dependence;
6. Allergic to sulfonamides or glibenclamide tablets;
7. The international normalized ratio was more than 1.4;
8. Renal insufficiency, history of dialysis treatment or serum creatinine more than 2.5 mg / dl;
9. Liver cirrhosis or severe liver dysfunction (ALT > 2.5 times the upper normal limit or total bilirubin > 1.5 times the upper normal limit);
10. He is taking bosentan tablets to treat pulmonary hypertension;
11. There was a history of glucose-6-phosphate dehydrogenase deficiency (faba bean disease);
12. The life expectancy is less than one year;
13. The gastrointestinal tract should not be used;
14. Pregnancy or lactation;
15. History of participating in other drug trials within 30 days;
16. There were clinical conditions that other researchers did not consider to meet the inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-10-19 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Serum neuron-specific enolase（NSE） | at 1st, 3rd,7th days after recruitment
  change of NSE serum concentrations after treatment
Change from Baseline Serum S100 β | at 1st, 3rd,7th days after recruitment
  change of S100B serum concentrations after treatment

SECONDARY OUTCOMES:
The proportion of modified Rankin score (0-2) | at 90 days
  The proportion of modified Rankin score (0-2)
The degree of brain edema | on the 3rd and 7th day after medication
  showed by brain CT
The incidence of delayed cerebral ischemia | up to 3 weeks
  The incidence of delayed cerebral ischemia
The incidence of hypoglycemia | up to 7 days
  The incidence of hypoglycemia
Intracranial pressure | up to 7 days
  if have

CONTACTS AND LOCATIONS:
Overall Officials: guangzhi shi, doctor, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lin Q, Zhou D, Ma J, Zhao J, Chen G, Wu L, Li T, Zhao S, Wen H, Yu H, Zhang S, Gao K, Yang R, Shi G. Efficacy and Safety of Early Treatment with Glibenclamide in Patients with Aneurysmal Subarachnoid Hemorrhage: A Randomized Controlled Trial. Neurocrit Care. 2024 Dec;41(3):828-839. doi: 10.1007/s12028-024-01999-z. Epub 2024 Aug 8. PMID 39117964